CLINICAL TRIAL: NCT04060290
Title: Real-world Study for the Safety of Albumin-Bound Paclitaxel in Malignant Tumors
Status: Completed | Type: Observational
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSPC-KAL-AE-01
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational study of this study, no interventions involved

SUMMARY:
This is a multi-center, Prospective, observational study，to evaluate the safety and influencing factors of albumin-bound paclitaxel in the real-world chinese population，and evaluate of the efficacy of albumin-bound paclitaxel in patients with malignant tumors and its impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* In patients with malignant tumor who have been treated with albumin-bound paclitaxel for the treatment.

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: malignant tumor
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage and severity of Participants With Adverse Events (AEs) | 28 days after the end of the last chemotherapy cycle
  percentage and CTC AE(v5.0) of AEs

SECONDARY OUTCOMES:
Objective response rate (ORR) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From signing informed consent，assessed up to end of study (up to approximately 24months)
  ORR is defined as the rate of CR or PR, as determined by IRC using RECIST v1.1 criteria.
evaluate patients' quality of life by the European Cancer Research and Treatment Tissue Cancer Quality Core Questionnaire EORTCQLQ-C30 | From signing informed consent，assessed up to end of study (up to approximately 24months)
  EORTC QLQC30 scale was used to score the quality of life before treatment, at each chemotherapy cycle, and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Study Director — Shiyao Group Ouyi Pharmaceutical Co., Ltd.
Locations (14):
- China (14):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Maanshan People's Hospital, Maanshan, Anhui
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Inner Mongolia Autonomous Region Cancer Hospital, Hohhot, Inner Mongolia
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hospital), Xi’an, Shanxi
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He F, Sun Y, Zhang W, Wu Q, Xu D, Bai Z, Hao Z, Feng W, Zhang K, Liu J, Dong M, Liu G, Li G. Safety and efficacy of generic nab-paclitaxel-based therapy in Chinese patients with malignant tumors in a real-world setting: a multicenter prospective observational study. Discov Oncol. 2024 Nov 26;15(1):712. doi: 10.1007/s12672-024-01609-6. PMID 39589666